CLINICAL TRIAL: NCT02263131
Title: Randomized, Double Blind, Active-controlled, Phase Ⅲ Study to Evaluate the Immunogenicity and Safety of 'Ilyang Flu Vaccine Pre-filled Syringe Inj.(Influenza Split Vaccine)' in Healthy Children Aged From 6 Months to < 18 Years.
Brief Title: Phase 3 Study to Evaluate the Immunogenicity and Safety of Inactivated Split Influenza Vaccine in Healthy Korea Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IY_IFEZ_CH_301
Record Dates: First submitted 2014-09-23; First posted 2014-10-13 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Influenza; Influenza vaccine; Split influenza vaccine; Seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IL-YANG PFS (Experimental): IL-YANG FLU Vaccine Prefilled Syringe INJ.
  Interventions: Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ.
- TIV PFS (Active Comparator): VAXIGRIP Prefilled Syringe INJ.
  Interventions: Biological: VAXIGRIP Prefilled Syringe INJ.

INTERVENTIONS:
Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ. — IL-YANG FLU Vaccine Prefilled Syringe INJ.0.5mL or 0.25mL
  Arms: IL-YANG PFS
Biological: VAXIGRIP Prefilled Syringe INJ. — VAXIGRIP Prefilled Syringe INJ.0.5mL or 0.25mL
  Arms: TIV PFS

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of IL-YANG Inactivated Split Influenza Vaccine (IL-YANG FLU Vaccine Prefilled Syringe INJ.) administered as a single intramuscular injection.

DETAILED DESCRIPTION:
This was a multi-center, randomized, double-blind, active-controlled study.

Before initiation of any protocol-specific activities, written informed consent was obtained from each patient and their legally acceptable representatives (consent of the legally acceptable representative was required for children younger than 10 years of age, and for the some sites, for children younger than 7 years of age). Subjects who met all of the eligibility criteria after screening assessments as specified in the protocol, were randomized into the test group or the comparator group in a ratio of 5 to 1 according to the pre-generated site-specific randomization table, and received a single dose or two doses of the study vaccine. The investigator performed the efficacy (immunogenicity) and safety assessments throughout the study. Efficacy data were collected at Visit 1 (prior to vaccination) and at the end-of-study visit for efficacy (immunogenicity) assessments, and for safety assessment, subjects and their legally acceptable representatives were instructed to record any treatment-emergent adverse event in Patient Diary cards.

For all randomized subjects, blood sample was obtained prior to vaccination, and the study vaccine 0.5mL or 0.25mL was administered to the deltoid muscle or anterolateral thigh muscle. For children aged from 6 months to <9 years of age who had not been previously exposed to influenza virus or had not previously received influenza vaccine, another dose of the study vaccine was administered 4 to 5 weeks after the first dose. Blood samples were collected 4 to 5 weeks after the last dose of the study drug for the assessment of antibody titer. All subjects were followed for 6 months after the last dose of the study drug for the safety assessments, and Month 6 follow-up visit was the end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged from 6 months to < 18 years
* Subjects were born after full term pregnancy (37 weeks)
* Voluntary written informed consent was obtained from the subject and the subject's legally acceptable representative (consent of legally acceptable representative was required for subjects younger than 10 years of age (and for subjects younger than 7 years of age for the some institutions)).

Exclusion Criteria:

* Subject with a known allergy to eggs, chicken, neomycin, gentamicin or any components of the study vaccine
* Subject who had received an influenza vaccine within the last 6 months
* Subject who has, or has a family history of, an immune system disorder including immune deficiency disease
* Subject with a history of Guillain-Barre syndrome
* Subject with Down's syndrome or cytogenetic disorders.
* Subject with severe chronic disease which in the investigator's opinion would not make the subject a good candidate for the clinical trial
* Subject with hemophilia or being treated with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection
* Subject who had an acute fever with body temperature > 38.0 Cº within 72 hours prior to administration of the study vaccine
* Subject who had previously received another vaccine within 28 days before administration of the study drug, or is scheduled to receive another vaccine during the study period.
* Subject who had received immunosuppressant or immune modifying drug within the last 3 months prior to administration of the study vaccine
* Subject who had previously received immunoglobulin or blood-derived products within the last 3 months prior to administration of the study vaccine, or is expecting to be treated with immunoglobulin or blood-derived products during the study.
* Subject who had participated in another experimental study within 30 days prior to administration of the study vaccine
* Subject with other clinically significant medical or psychological condition who in the investigator's opinion would not be suitable for the study.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 416 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Han Kang, MD.PhD, Principal Investigator — Seoul St. Mary's Hospital, The Catholic University of Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IL-YANG PFS | TIV PFS
Started | 347 | 69
Completed | 337 | 68
Not Completed | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IL-YANG PFS | TIV PFS | Total
Number analyzed (Participants) | 347 | 69 | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.83 (4.87) | 7.45 (5.01) | 7.77 (4.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 34 | 225
  Male | 156 | 35 | 191

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Healthy Children Aged From 6 Months to <18 Years With Seroconversion
Description: Seroconversion is defined as follows. (Case 1) A pre-vaccination (Day 0) HI antibody titer < 1:10 and a post-vaccination (Day 28) HI antibody titer ≥ 1: 40. or (Case 2) a pre-vaccination (Day 0) HI antibody titer ≥ 1:10 and a minimum four-fold rise in post-vaccination (Day 28) HI antibody titer.
Time Frame: up to Day28(+7)
Population: Whole participant
Measure: Number; unit: percentage of paticipants
Arm/Group | IL-YANG PFS | TIV PFS
Number analyzed (Participants) | 337 | 68
percentage of paticipants
  Strain H1N1 | 62.02 | 76.81
  Strain H3N2 | 53.41 | 57.35
  Strain B | 54.90 | 66.18

2. Primary Outcome: Percentage of Subjects Achieving Seroconversion for HI Antibody After Administration of the Study Vaccine Depending of the Number of Vaccination
Description: Seroconversion: a pre-vaccination (Day 0) hemagglutination-inhibition (HI) antibody titer < 1:10 and a post-vaccination (last vaccination + Day 28) HI antibody titer ≥ 1: 40 (Case 1), or a pre-vaccination (Day 0) HI antibody titer ≥ 1:10 and a minimum four-fold rise in post-vaccination (last vaccination + Day 28) HI antibody titer (Case 2),
Time Frame: up to Day28(+7)
Population: This is because the results showed that the seroconversion rate of HI antibody varies depending on the number of vaccination.
Measure: Number; unit: percentage of participants
Arm/Group | IL-YANG PFS | TIV PFS
Number analyzed (Participants) | 337 | 68
percentage of participants
  Strain H1N1(1st): number analyzed (Participants) | 308 | 62
  Strain H1N1(1st) | 60.06 | 54.84
  Strain H1N1(2nd): number analyzed (Participants) | 29 | 6
  Strain H1N1(2nd) | 82.76 | 66.67
  Strain H3N2(1st): number analyzed (Participants) | 308 | 62
  Strain H3N2(1st) | 53.41 | 56.45
  Strain H3N2(2nd): number analyzed (Participants) | 29 | 6
  Strain H3N2(2nd) | 75.86 | 66.67
  Strain B(1st): number analyzed (Participants) | 308 | 62
  Strain B(1st) | 54.22 | 66.13
  Strain B(2nd): number analyzed (Participants) | 29 | 6
  Strain B(2nd) | 62.07 | 66.67

3. Primary Outcome: Seroprotection Rate for HI Antibody
Description: Percentage of Participants With Healthy Children Aged From 6 Months to <18 Years With Seroprotection
Time Frame: up to Day28(+7)
Population: Whole participant
Measure: Number; unit: percentage of paticipants
Arm/Group | IL-YANG PFS | TIV PFS
Number analyzed (Participants) | 337 | 68
percentage of paticipants
  Strain H1N1 | 94.96 | 89.71
  Strain H3N2 | 93.77 | 91.18
  Strain B | 95.25 | 95.59

4. Primary Outcome: Seroprotection Rate of HI Antibody
Description: Percentage of subjects achieving seroprotection for HI antibody after administration of the study vaccine depending of the number of vaccination
Time Frame: up to Day28(+7)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | IL-YANG PFS | TIV PFS
Number analyzed (Participants) | 337 | 68
percentage of participants
  Strain H1N1(1st): number analyzed (Participants) | 308 | 62
  Strain H1N1(1st) | 96.10 | 91.94
  Strain H1N1(2nd): number analyzed (Participants) | 29 | 6
  Strain H1N1(2nd) | 82.76 | 66.67
  Strain H3N2(1st): number analyzed (Participants) | 308 | 62
  Strain H3N2(1st) | 95.45 | 93.55
  Strain H3N2(2nd): number analyzed (Participants) | 29 | 6
  Strain H3N2(2nd) | 75.86 | 66.67
  Strain B(1st): number analyzed (Participants) | 308 | 62
  Strain B(1st) | 96.75 | 96.77
  Strain B(2nd): number analyzed (Participants) | 29 | 6
  Strain B(2nd) | 79.31 | 83.33

5. Secondary Outcome: Geometric Mean Titer* (GMT) of HI Antibody
Description: Geometric Mean Titer (GMT), as measured by pre-vaccination (Day 0) HI antibody titer and post-vaccination (vaccination + 28 days) HI antibody titer.
Time Frame: Day28(+7)
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | IL-YANG PFS | TIV PFS
Number analyzed (Participants) | 337 | 68
Titer
  Strain H1N1(pre) | 24.40 [21.99 to 27.07] | 24.80 [19.76 to 31.12]
  Strain H1N1(post) | 111.40 [101.52 to 122.25] | 88.45 [70.33 to 111.24]
  Strain H3N2(pre) | 31.85 [28.47 to 35.63] | 30.00 [22.59 to 39.84]
  Strain H3N2(post) | 110.60 [100.93 to 121.19] | 104.92 [82.25 to 133.84]
  Strain B(pre) | 36.22 [32.63 to 40.21] | 39.44 [31.96 to 48.66]
  Strain B(post) | 130.53 [117.98 to 144.41] | 151.70 [119.0 to 192.90]

6. Secondary Outcome: GMR of HI Antibody Titer Before Vaccination and After Vaccination
Description: Geometric Mean Ratio (GMR), as measured by pre-vaccination (Day 0) HI antibody titer and post-vaccination (vaccination + 28 days) HI antibody titer.
Time Frame: Day28(+7)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio of GMT titer
Arm/Group | IL-YANG PFS | TIV PFS
Number analyzed (Participants) | 337 | 68
Ratio of GMT titer
  Strain H1N1 | 4.57 [4.11 to 5.08] | 3.57 [2.79 to 4.57]
  Strain H3N2 | 3.47 [3.16 to 3.82] | 3.50 [2.77 to 4.42]
  Strain B | 3.60 [3.26 to 3.98] | 3.85 [3.01 to 4.92]

7. Secondary Outcome: Number of Subjects With a Pre-vaccination (Day 0) HI Antibody Titer < 1:40, Minimum Four-fold Rise in Post-vaccination (Day 28) HI Antibody Titer
Time Frame: Day28(+7)
Population: Number of subjects whose HI antibody titer increased minimum four-fold on day 28 after vaccination
Measure: Number; unit: percentage of participants
Arm/Group | IL-YANG PFS | TIV PFS
Number analyzed (Participants) | 54 | 16
percentage of participants
  Strain H1N1: number analyzed (Participants) | 17 | 7
  Strain H1N1 | 35.29 | 28.57
  Strain H3N2: number analyzed (Participants) | 21 | 6
  Strain H3N2 | 61.90 | 50.00
  Strain B: number analyzed (Participants) | 16 | 3
  Strain B | 18.75 | 0.00

ADVERSE EVENTS:
Arm/Group | IL-YANG PFS | TIV PFS
Serious Adverse Events (participants affected / at risk) | 8/347 | 0/69
Other Adverse Events (participants affected / at risk) | 185/347 | 41/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IL-YANG PFS (N=347) | TIV PFS (N=69)
Febrile convulsion (Nervous system disorders) | 1 | 0
Kawasaki's disease (Vascular disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IL-YANG PFS (N=347) | TIV PFS (N=69)
Pain (Skin and subcutaneous tissue disorders) | 120 | 25
Tenderness (Skin and subcutaneous tissue disorders) | 168 | 35
Redness (Skin and subcutaneous tissue disorders) | 48 | 5
Swelling (Skin and subcutaneous tissue disorders) | 19 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No